CLINICAL TRIAL: NCT06133049
Title: Zeposia (Ozanimod) Pregnancy Study: A Retrospective Observational Study on the Safety of Ozanimod Exposure in Pregnant Women and Their Offspring
Brief Title: A Study to Evaluate the Safety of Ozanimod Exposure During Pregnancy in Women With Multiple Sclerosis and Their Infants
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM047-002
Record Dates: First submitted 2023-10-18; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ozanimod

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ozanimod exposed
  Interventions: Drug: Ozanimod
- Other DMT exposed
  Interventions: Drug: Select DMTs other than ozanimod
- Not DMT exposed
  Interventions: Drug: No DMTs

INTERVENTIONS:
Drug: Ozanimod — Women with MS who were exposed to ozanimod during pregnancy
  Groups: Ozanimod exposed
Drug: Select DMTs other than ozanimod — Women with MS exposed to select DMTs other than ozanimod during pregnancy
  Groups: Other DMT exposed
Drug: No DMTs — Women with MS not exposed to any DMTs during pregnancy
  Groups: Not DMT exposed

SUMMARY:
The purpose of this retrospective observational cohort study is to assess pregnancy and infant outcomes in three groups: the first is women with multiple sclerosis (MS) who were exposed to ozanimod during pregnancy; the second is women with MS exposed to select other disease-modifying therapies (DMTs) during pregnancy; the third is women with MS not exposed to any DMTs during pregnancy. This study will use data from a large US healthcare claims database.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 49 years at date of conception
* Date of conception between April 1, 2020 and July 31, 2030

Exclusion Criteria:

* Pregnancies exposed to any known teratogens and the exposure falls within the period of 5 half-lives prior to the estimated date of conception through the end of the first trimester (assessed via the presence of national drug codes or medical procedure codes)
* Exposure to the DMTs fingolimod, siponimod, mitoxantrone, and teriflunomide within a period of 5 half-lives prior to the estimated date of conception through the end of the first trimester

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant adult women with MS with an estimated date of conception between April 1, 2020 and July 31, 2030
Sampling Method: Non-Probability Sample
Enrollment: 2961 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2031-03-31 (Estimated); Study Completion 2031-08-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of major congenital malformations among infants | Up to 11 years
  Prevalence of major congenital malformations among infants born to women with MS exposed to ozanimod during the first trimester, and to compare this to the prevalence among each of the two comparator groups of pregnant women (other DMT exposed or NO DMT exposed)

SECONDARY OUTCOMES:
Number of spontaneous abortions | Up to 11 years
Number of preterm births | Up to 11 years
Number of stillbirths | Up to 11 years
Number of participants with pre-eclampsia | Up to 11 years
Number of participants with eclampsia | Up to 11 years
Number of infants small for gestational age | Up to 11 years
Number of serious or opportunistic infections in liveborn infants up to one year of age | Up to 11 years
Number of infant postnatal growth deficiencies | Up to 11 years
Number of infant developmental deficiencies | Up to 11 years
Number of neonatal hospitalizations | Up to 11 years
Number of infant deaths | Up to 11 years
Number of neonatal deaths | Up to 11 years
Number of perinatal deaths | Up to 11 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- OptumInsight Life Sciences Inc, Eden Prairie, Minnesota, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html